CLINICAL TRIAL: NCT02992639
Title: Weight Loss Effect on Circulating Levels of Liver Enzymes in Overweight Subjects With High Visceral Fat Area: 12-week Randomized Controlled Trial
Brief Title: Weight Loss Effect on Circulating Liver Enzymes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VFA_liver enzyme
Record Dates: First submitted 2016-12-11; First posted 2016-12-14 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-01

CONDITIONS: Visceral Fat; Liver Dysfunction
Keywords: High visceral fat; Liver enzymes; Aminotransferase; Mild calorie restriction
MeSH Terms: conditions — Liver Diseases | interventions — Control Groups

ARMS (2):
- Control group (Placebo Comparator): No calorie restriction group
  Interventions: Behavioral: Control group
- Weight loss group (Experimental): Mild calorie restriction group (300kcal/day intake reduction)
  Interventions: Behavioral: Weight loss group

INTERVENTIONS:
Behavioral: Control group — The participants who included in control group did not receive any treatment.
  Arms: Control group
Behavioral: Weight loss group — The participants who included in weight loss group followed a 12-week weight loss program consisting of a 300 kcal/day reduction of thier usual caloric intakes
  Arms: Weight loss group

SUMMARY:
To investigate weight loss effect with mild calorie restriction on circulating levels of liver enzymes in nondiabetic and overweight subjects with high visceral fat area [visceral fat area (VFA) at L4 ≥ 100 cm²].

DETAILED DESCRIPTION:
A 12-week randomized, placebo-controlled study was conducted on 80 nondiabetic and overweight subjects with high VFA. The participants divided into two groups: 12-week mild calorie restriction (a 300 kcal/day intake reduction, n=40) or no treatment (control, n=40). The randomization was according to computer-generated block randomization (placebo:test = 1:1). Before and after intervention period, venous blood samples were obtained from the subjects, and biochemical parameters including circulating liver enzymes were measured.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent
* 20-60 years old
* Males and females
* Overweight (25.0 kg/m²≤ BMI <30 kg/m²)
* Absence of pregnancy or breast-feeding
* Stable body weight (body weight change <1kg for 3 months before screening)
* High visceral fat (VFA) at L4 (VFA at L4 ≥100 cm²)
* Without hypertension, type 2 diabetes, cardiovascular disease, or thyroid disease
* No use medication affecting body weight, energy expenditure, or glucose control for the last 6 months

Exclusion Criteria:

* Prior history of Cushing syndrome or malignancy
* Prior history of liver disease including chronic viral hepatitis, autoimmune hepatitis, primary biliary cirrhosis, or drug-induced liver disease
* Excess alcohol intake (based on WHO standard)
* History of intentional reduction in weight in the preceding 6 months

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2015-06; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Visceral fat area at L4 (CT) | At baseline
Visceral fat area at L4 (CT) | At 12-week follow-up
Change from baseline visceral fat area at L4 at 12-week (CT) | At baseline and 12-week follow-up
Serum fatty acid levels (Relative peak area) | At baseline
Serum fatty acid levels (Relative peak area) | At 12-week follow-up

SECONDARY OUTCOMES:
Fat percentage (DEXA) | At baseline
Fat percentage (DEXA) | At 12-week follow-up
Change from baseline fat percentage at 12-week (DEXA) | At baseline and 12-week follow-up
Fat mass (DEXA) | At baseline
Fat mass (DEXA) | At 12-week follow-up
Change from baseline fat mass at 12-week (DEXA) | At baseline and 12-week follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Jong Ho Lee, PhD, Principal Investigator — Yonsei University
Locations (1):
- Yonsei University, Seoul, South Korea

REFERENCES:
- [Derived] Lee YJ, Lee A, Yoo HJ, Kim M, Kim M, Jee SH, Shin DY, Lee JH. Effect of weight loss on circulating fatty acid profiles in overweight subjects with high visceral fat area: a 12-week randomized controlled trial. Nutr J. 2018 Feb 22;17(1):28. doi: 10.1186/s12937-018-0323-4. PMID 29471812